CLINICAL TRIAL: NCT05097469
Title: Randomized, Double-blind, Sham-controlled Clinical Trial for Evaluating the Efficacy of Fractional Carbon Dioxide Laser in the Treatment of Female Sexual Dysfunction.
Brief Title: Carbon Dioxide Acupulse Laser Treatment Versus Sham Treatment and Sexual Dysfunction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0290-20-RMB
Record Dates: First submitted 2021-10-04; First posted 2021-10-28 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Lasers, Gas

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser treatment (Active Comparator): Carbon dioxide laser treatment
  Interventions: Device: Carbon dioxide laser
- Sham treatment (Sham Comparator): Sham laser treatment
  Interventions: Device: Sham laser treatment

INTERVENTIONS:
Device: Carbon dioxide laser — 3 consecutive sessions of carbon dioxide laser treatment
  Arms: Laser treatment
Device: Sham laser treatment — 3 consecutive sessions of sham laser treatment
  Arms: Sham treatment

SUMMARY:
The study is intended to assess the safety and efficacy of Carbon dioxide AcuPulse laser treatment in patients with sexual dysfunction. Eligible subjects will be randomized to either receive 3 laser or 3 sham treatment sessions, 4 weeks apart and 3 follow up visits 3, 6 and 12 months following the last treatment.

DETAILED DESCRIPTION:
Following a screening visit, eligible subjects will be enrolled into the study. Subjects will be randomized into either laser treatment or sham treatment. Each subject will receive 3 treatments 4 weeks apart and 3 follow up visits, at 3, 6 and 12 months following the last treatment.

Further demographic information and patient history will be obtained from the subjects' electronic files.

ELIGIBILITY:
Inclusion Criteria:

* Negative urine analysis.
* Normal Pap smear test from the recent 3 years.
* No previous gynecological laser treatments.
* Able and willing to comply with the treatment/follow-up schedule and requirements.

Exclusion Criteria:

* Active genital infection.
* Subject presenting abnormal Pap result from the last three years.
* Recurring urinary tract infection or recurring infection of genital herpes or candida (> 2 episodes in the recent year).
* Transvaginal mesh implant.
* Serious systemic disease or any chronic condition that could interfere with study compliance.
* Any vaginal bleeding of unknown reason.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Enrollment: 120 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Vaginal health index | From treatment up to 12 months post treatment
  Change in total and specific vaginal health index scores

SECONDARY OUTCOMES:
Female sexual function index | From treatment up to 12 months post treatment
  Change in total and specific female sexual function index questionnaire scores
Sexual intercourse | From treatment up to 12 months post treatment
  Change in monthly sexual intercourse rate

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam healthcare campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No